CLINICAL TRIAL: NCT02624583
Title: Effects of Ramadan Fasting on Clopidogrel Resistance in Patients at High Cardiovascular Risk. An Observational Study
Brief Title: Effects of RF on Clopidogrel Resistance in Patients at High Cardiovascular Risk
Acronym: RFeCloR
Status: Completed | Type: Observational
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, Professor, University of Monastir
Other Study IDs: 08/2015
Record Dates: First submitted 2015-12-03; First posted 2015-12-08 (Estimated); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Coronary Artery Disease; Diabetes Mellitus
Keywords: Fasting; Clopidogrel
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus; Fasting

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Venous blood samples were collected from the enrolled participants. Blood samples were analyzed for hemoglobin, hematocrit, platelet cell count, Prothrombin time, activated partial thromboplastin time, and clopidogrel effect on P2Y12 receptor by optical turbidimetry (expressed as P2Y12 reaction units (PRU)).
Oversight: Data Monitoring Committee: No

SUMMARY:
Ramadan fasting (RF) has been shown to be associated with vascular and metabolic disorders including glycemic control and lipid profile. It may also alter pharmacologic properties of some medications. Many patients with coronary artery disease (CAD) and under Clopidogrel insist to observe the fasting and taking the risk of altering the pharmacologic proprieties of this drug.

The aim of this study is to assess the effects of RF on clopidogrel resistance in patients at high cardiovascular risk with particular interest to patients with Diabetes Mellitus (DM).

DETAILED DESCRIPTION:
The study involved three separate assessment visits in each year: 1) the last week before Ramadan (Pre-R) which represented the baseline period; 2) the last week of Ramadan (R); 3) and during the last week of the month following Ramadan(Post-R). Each patient served as his own control and was required to take the prescribed clopidogrel dose daily and chart the intake in a dosing diary. The duration of fasting was approximately 12 h from sunrise to sunset(the time of abstinence from food) during a 30 day period. The assessment in each of the three visits involved clinical exam and blood sampling for hematologic and metabolic tests

Body weight and height were performed by a well-trained staff member. Weight was measured while the subjects were minimally clothed without shoes using digital scales and recorded to the nearest 0.1 kg. Body Mass Index (BMI) was calculated as body weight (kg) divided by squared height in meters (m2). Physical examination was carried out in all participants including systolic (SBP), diastolic (DBP) blood pressure, and heart rate. The visit is completed by a questionnaire on diet beginning 2 days before the blood sampling. No special nutritional regimen was applied to the participants during the study. All subjects were encouraged to continue their usual lifestyle and activities.

The rate of hypoglycemic (symptomatic and non-symptomatic) and hyperglycemic episodes requiring emergency department (ED) admission was recorded within the three periods of the study. Hypoglycemia was defined as blood glucose <3.5 mmol/l. Compliance to current treatment (clopidogrel, oral hypoglycemic agents,statins...) was assessed by the attending physician based on interview and pill count. Venous blood samples were collected from the enrolled participants during the three time points. The time of blood sampling in the study was 9-10 a.m., at which all participants were fast. For the purpose of the study,we asked our patients to take clopidogrel treatment as late as possible.

As Ramadan month during the study period has coincided with summer season,clopidogrel was generally taken between midnight and1 am. We added this detail in the paper..

ELIGIBILITY:
Inclusion Criteria:

* aged more than 40 years old.
* having at least two cardiovascular risk factors according to Framingham classification.
* patients willing to fast ramadan and taking clopidogrel therapy for at least six months prior to inclusion.

Exclusion Criteria:

* patients under 40 years.
* patients with unstable diabetes.
* repeated hypoglycemic episodes
* patients with severe uncontrolled hypertension (higher arterial blood pressure than 179/109 mmHg despite antihypertensive treatment)
* acute coronary syndrome within the past year prior to enrollment
* current or previous (14 days) use of glycoprotein IIb/IIIa
* severe cardiovascular and cerebrovascular disease
* inability to give informed consent
* baseline platelet count < 100x103/ml
* current use of antidepressants
* serum creatinine levels higher than 1.4 mg/dL for women and 1.5 mg/dL for men
* hepatic function tests at least 2.5 times higher than normal levels
* terminal disease with a <1 year expected mortality

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were screened in outpatient clinics (cardiology, endocrinology, internal medicine, family medicine) when they presented for scheduled follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2010-06 (Actual); Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Changes in platelet reactivity between the three time points | the last week before Ramadan (Pre-R); the last week of Ramadan (R); and during the last week of the month following Ramadan (Post-R)
  the platelet reactivity to clopidogrel is assessed by the 'Verify Now P2Y12' point-of-care assay .
  Results are reported as P2Y12 reaction units (PRU); the lower the PRU value, the higher the platelet aggregation inhibition by clopidogrel.
  High platelet reactivity after clopidogrel (clopidogrel resistance) was defined at two cutoff values (PRU≥235 and ≥ 208).

SECONDARY OUTCOMES:
Changes in the glycemic profile between the three time points | the last week before Ramadan (Pre-R); the last week of Ramadan (R); and during the last week of the month following Ramadan (Post-R)
  An automated analyzer (Beckman Coulter DXC 600, UK) measured the concentrations of biochemical parameters using the appropriate reagents.
  Glucose concentrations are measured by an enzymatic colorimetric method and expressed in mmol/l.
Changes in the lipid profile between the three time points | the last week before Ramadan (Pre-R); the last week of Ramadan (R); and during the last week of the month following Ramadan (Post-R)
  An automated analyzer (Beckman Coulter DXC 600, UK) measured the concentrations of biochemical parameters using the appropriate reagents.
  The total cholesterol (TC) and triglycerides (TG) were determined using an enzymatic colorimetric method. High-density lipoprotein cholesterol (HDL-C) concentrations were determined by immuno-inhibition. Low-density lipoprotein cholesterol (LDL-C) was calculated using the Friedewald formula: LDL-C (mmol/L) =TC - HDL-C - TG: 2.2.

CONTACTS AND LOCATIONS:
Overall Officials: Semir Nouira, Professor, Principal Investigator — University of Monastir
Locations (2):
- Tunisia (2):
  - Emergency department of university hospital Fattouma Bourguiba of Monastir Monastir, Monastir Tunisia, Monastir
  - Fattouma Bourguiba University Hospital, Monastir